CLINICAL TRIAL: NCT00829556
Title: Single-Center, Randomized Trial to Study the Efficacy of InteguSeal for Surgical Skin Preparation in Patients Undergoing
Brief Title: Efficacy of InteguSeal for Surgical Skin Preparation in Patients Undergoing Total Joint Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: Kimberly-Clark Corporation (Industry)
Responsible Party: Javad Parvizi, MD, FRCS, Rothman Institute Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RIFJPAR 08-01
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Prosthetic Joint Infection; Surgical Skin Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Device: Integuseal
- 2 (No Intervention): Standard Surgical skin preparation

INTERVENTIONS:
Device: Integuseal
  Arms: 1

SUMMARY:
This study is being conducted to investigate the potential benefits of using a special type of fluid that can be applied to the skin (Integuseal) in addition to standard surgical skin preparation in patients undergoing total hip replacement (THA) or total knee replacement (TKA). Integuseal is supposed to lock down the skin bacteria and reduce skin infection and other problems. This study will investigate whether Integuseal is effective in reducing persistent wound drainage when used in addition to standard surgical skin preparation for total hip arthroplasty (THA) or total knee replacement (TKA).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able and willing to provide informed consent;
2. Male and non-pregnant, non-lactating, female subjects who are willing to practice effective means of contraception or postmenopausal/surgically sterilized female subjects, between the ages of 18-80 years old, of any ethnic origin.
3. Subjects deemed able to comply with study schedule visits, procedures and medications as specified by the protocol.
4. Subjects undergoing elective THA or TKA procedures.
5. Subjects in satisfactory health as determined by the investigator on the basis of medical history and physical examination.

Exclusion Criteria:

1. Subjects undergoing revision, hemiarthroplasty, or bilateral THA or TKA
2. Subjects undergoing non-elective THA or TKA procedures.
3. Pregnant or lactating females or females of childbearing potential not practicing an effective method of contraception.
4. Subjects with known allergies to iodine and/or chlorhexidine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study will be to determine the incidence of postoperative wound drainage during hospital stay when adding Integuseal to the normal surgical skin preparation. | Total joint replacement to discharge from hospital

SECONDARY OUTCOMES:
To evaluate the effect of using Integuseal on the length of hospital stay after THA or TKA. | Total joint replacement to discharge from hospital
To evaluate the effect of using Integuseal on the incidence of surgical site infection (SSI). | 6 weeks
To evaluate the effect of using Integuseal on the incidence of revision or re-admission after undergoing THA or TKA | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Javad Parvizi, MD, FRCS, Principal Investigator — Rothman Institute Orthopaedics
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States